CLINICAL TRIAL: NCT02935348
Title: Feasibility of Using Whole Body PET-MRI to Stage and Restage Paediatric and Adolescent Hodgkin Lymphoma - a Pilot Study
Brief Title: Whole Body PET-MRI in Paediatric and Adolescent Lymphoma
Acronym: PET/MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 13/0268
Record Dates: First submitted 2015-12-03; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2015-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Whole Body MRI — Routine whole body clinical MRI will be performed according to current clinical standard of care. Axial and coronal imaging from the maxilla to proximal femurs will be performed using a combination of T1 and T2 weighted sequences, with and without gadolinium administration.

SUMMARY:
Children and adolescents with Hodgkin lymphoma currently undergo multiple investigations including a separate PET and MRI scans during their treatment.

Investigators want to investigate if a combined PET-MRI scan could give the same information.

Children who join our study will have an extra scan twice during their treatment

DETAILED DESCRIPTION:
Children and adolescents with Hodgkin lymphoma currently undergo multiple investigations including a separate PET and MRI scans during their treatment.

Investigators want to investigate if a combined PET-MRI scan could give the same information.

Children who join our study will have an extra scan twice during their treatment

Routine whole body clinical MRI will be performed according to current clinical standard of care. Axial and coronal imaging from the maxilla to proximal femurs will be performed using a combination of T1 and T2 weighted sequences, with and without gadolinium administration.

ELIGIBILITY:
Inclusion Criteria:

1. Suspected or histologically confirmed Hodgkin lymphoma
2. Male or female participants
3. Age 0-20 years inclusive
4. Entered into the EuroNet PHL-C1 trial, LP1 trial or successor Euronet trials, including Euronet PHL C2 due to open from 2013 onwards or planned to receive chemotherapy regimens of said trials without being formally entered into the trial.
5. Participant/Guardian/Parental written informed consent

Exclusion Criteria:

1. Participants with contraindications to MRI (including cardiac pacemakers or non-MRI compatible intracranial vascular clips)
2. Participants who are pregnant or nursing

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Childhood and adolescent cases of clinically suspected or histologically confirmed Hodgkin Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The investigator will determine the technical feasibility of performing functional co-registered combined PET-MRI in this patient group using diffusion-weighted MR imaging. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Humphries, Principal Investigator — UCL
Locations (1):
- Centre for Medical Imaging, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes